CLINICAL TRIAL: NCT03304054
Title: A Randomized, Placebo-control, Parallel Group Study to Evaluate the Effect of Amifampridine Phosphate in Patients With MuSK Antibody Positive Myasthenia Gravis, and a Sample of AChR Antibody Positive Myasthenia Gravis Patients
Brief Title: Study to Evaluate Amifampridine Phosphate in Patients With MuSK-MG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSK-002
Record Dates: First submitted 2017-09-28; First posted 2017-10-06 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2021-07

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: MuSK antibody positive
MeSH Terms: conditions — Myasthenia Gravis | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- amifamapridine phosphate tablets (Experimental)
  Interventions: Drug: Amifampridine Phosphate
- placebo tablets (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Amifampridine Phosphate — tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day
  Arms: amifamapridine phosphate tablets
Drug: Placebo Oral Tablet — tablets matching amifampridine phosphate, 3 to 4 times a day
  Arms: placebo tablets

SUMMARY:
Efficacy and safety of amifampridine phosphate in improving the activities of daily living for patients with antibody positive MuSK myasthenia gravis.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel group study is designed to evaluate the safety, tolerability and efficacy of amifampridine phosphate in patients with MuSK-MG. In addition, a sample of AChR-MG patients will be assess for efficacy and safety of amifampridine phosphate. Planned duration of participation for each patient is at least 38 days, excluding the screening period. Eligible patients will be titrated to an efficacious dose of amifampridine phosphate and those who demonstrate improvement will be randomized to either placebo or amifampridine, in a double-blind fashion, for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.
2. Male or female ≥18 years of age.
3. Positive serologic test for anti-MuSK antibodies or anti-AChR antibodies as confirmed at Screening or by previous antibody test, with report available.
4. Confirmatory EMG or EMG report.
5. Myasthenia Gravis Foundation of America (MGFA) Class II to IV at Screening.
6. MG-ADL score of ≥6 at Screening, with more than 50% of this score attributed to non-ocular items.
7. Patients receiving steroids or pyridostigmine should not have any modification of drug regimen during the month before Screening.
8. Female patients of childbearing potential must have a negative pregnancy test (serum human chorionic gonadotropin [HCG] at screening); and must practice an effective, reliable contraceptive regimen during the study and for up to 30 days following discontinuation of treatment.
9. Ability to participate in the study based on overall health of the patient and disease prognosis, as applicable, in the opinion of the Investigator; and able to comply with all requirements of the protocol, including completion of study questionnaires.

Exclusion Criteria:

1. Epilepsy and currently on medication.
2. Concomitant use of medicinal products with a known potential to cause QTc prolongation.
3. Patients with long QT syndromes.
4. History of thymectomy within 12 months before Screening.
5. An electrocardiogram (ECG) within 6 months before starting treatment that shows clinically significant abnormalities, in the opinion of the Investigator.
6. Breastfeeding or pregnant at Screening or planning to become pregnant at any time during the study.
7. Patients receiving immunomodulatory treatment (e.g. plasma exchange [PE], therapeutic plasma exchange [TPE], intravenous immunoglobulin G [IVIG]) should not have any treatment in the previous 4 weeks prior to Randomization or at any time during the study.
8. Use of rituximab or other similar biologic medications for immunomodulation within 6 months prior to Screening.
9. Treatment with an investigational drug (other than amifampridine) or device within 30 days before Screening or while participating in this study.
10. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confound the assessment of the patient.
11. History of drug allergy to any pyridine-containing substances or any amifampridine excipient(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Mantegazza, MD, Principal Investigator — Carlo Besta Neurologic Institute
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Univerity of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 18 April 2018 - 24 April 2020 at 26 sites in the United States and Europe.
Pre-assignment Details: A screening visit was conducted to ensure that each patient met inclusion/exclusion criteria. Those patients successfully completing screening had procedures/assessments conducted at the start of the Run-in period (Day 1, before starting study medication) and during run-in, until stable dose and frequency of amifampridine is established for at least 7 days, and at least a 2-point improvement in MG-ADL score was achieved from the start of Run-in to be eligible for randomization (Day 0).
Groups:
- Amifampridine Phosphate - MuSK: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day
  MuSK - patients diagnosed with MuSK-MG
- Amifampridine Phosphate - AChR-MG: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day
  AChR-MG- patients diagnosed with AChR-MG
- Placebo - MuSk: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
  MuSK - patients diagnosed with MuSK-MG
- Placebo - AChR-MG: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
  AChR-MG- patients diagnosed with AChR-MG
- Amifampridine Phosphate Only - MuSK: Patients receiving amifampridine during the open-label run-in period but were not randomized for the crossover portion of the study and diagnosed with MuSK-MG.
- Amifampridine Phosphate Only- AChR-MG: Patients receiving amifampridine during the open-label run-in period but were not randomized for the crossover portion of the study and diagnosed with AChR-MG.
Period: Overall Study
Arm/Group | Amifampridine Phosphate - MuSK | Amifampridine Phosphate - AChR-MG | Placebo - MuSk | Placebo - AChR-MG | Amifampridine Phosphate Only - MuSK | Amifampridine Phosphate Only- AChR-MG
Started | 27 | 7 | 28 | 8 | 17 | 6
Completed | 27 | 7 | 27 | 8 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 17 | 6

BASELINE CHARACTERISTICS:
Population: The analysis of baseline characteristics included all patients in the Safety population, who are those patients who enrolled and received at least one dose of amifampridine. Patients who began the run-in period belong to the Safety population whether they were randomized to treatment or not.
Groups:
- Placebo: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
- Amifampridine Phosphate Only: Patients receiving Amifampridine during the open-label Run-in period but were not randomized for the crossover portion of the study.
- Total: Total of all reporting groups
Arm/Group | Amifampridine Phosphate | Placebo | Amifampridine Phosphate Only | Total
Number analyzed (Participants) | 34 | 36 | 16 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (14.92) | 53.5 (12.61) | 45.9 (11.31) | 51.9 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 14 | 66
  Male | 10 | 8 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 15 | 18
  Not Hispanic or Latino | 33 | 34 | 1 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 7
  White | 31 | 34 | 13 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 84.6 (21.11) | 84.3 (27.27) | 76.1 (32.28) | 82.9 (25.96)
Height [Mean (Standard Deviation); unit: cm] | 164.7 (7.64) | 163.5 (10.75) | 163.6 (7.37) | 164.0 (8.99)

OUTCOME MEASURES:

1. Primary Outcome: Myasthenia Gravis-Activities of Daily Living (MG-ADL) Summary by Time Point and Myasthenia Gravis Type: Wilcoxon-Mann-Whitney Rank Sum Test Results
Description: Myasthenia Gravis-Activities of Daily Living (MG-ADL) is a self-report scale to assess the patient's MG symptoms and functional performance of activities of daily living. The eight items are scored on a scale of 0-3 with 3 representing the most severe symptoms or impaired performance and 0 representing no symptoms or impaired performance. Each item was assessed by the patient at the last day (Day 0) of the Run-in period and at the post-treatment visit. The post-treatment result will be the result obtained on Day 10. If the patient discontinued treatment early, the post-treatment result may be obtained at an earlier time point. The total MG-ADL score was calculated as the sum of each item score, with a maximum score of 24 (most severe symptoms/impairment) and minimum score of 0 (least severe symptoms/impairment). The change from baseline (CFB) at Day 10 was assessed. A Wilcoxon-Mann-Whitney Rank Sum Test of equality of change from baseline distributions between subjects diagnos
Time Frame: Last day (Day 0) of the Run-in period and at the post-treatment visit (i.e., day 10 or the time point at which a patient discontinued treatment early).
Population: The analysis of primary outcome data was based on the Full Analysis Set population, which included all randomized patients who received at least one dose of study medication (amifampridine or placebo post randomization) and had at least one post-treatment efficacy assessment. Patients who discontinued with no post-randomization data (no Day 0 and no Day 10 data) were excluded from all efficacy analyses but were included in the safety analyses.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Amifampridine Phosphate - MuSK: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day
  Patients randomized to receive Amifampridine and diagnosed with MuSK-MG.
- Placebo - MuSK: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
  Patients randomized to receive Placebo and diagnosed with MuSK-MG.
- Amifampridine Phosphate - AChR: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day
  Patients randomized to receive Amifampridine and diagnosed with AChR-MG.
- Placebo - AChR: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
  Patients randomized to receive Placebo and diagnosed with AChR-MG.
Arm/Group | Amifampridine Phosphate - MuSK | Placebo - MuSK | Amifampridine Phosphate - AChR | Placebo - AChR
Number analyzed (Participants) | 27 | 28 | 7 | 8
Score on a Scale
  Baseline (Day 0) MG-ADL Total Raw Score | 4.96 (2.915) | 3.86 (2.103) | 6.14 (3.388) | 7.00 (4.175)
  Post-Baseline(Day 10 or time at which a patient discontinued treatment) MG-ADL Total Raw Score | 6.00 (3.658) | 6.11 (3.19) | 4.71 (3.147) | 10.38 (3.583)
  CFB MG-ADL Total Score | 1.04 (2.980) | 2.25 (3.658) | -1.43 (2.225) | 3.38 (2.825)
Statistical Analysis 1: Comparison: Amifampridine Phosphate - MuSK vs Placebo - MuSK vs Amifampridine Phosphate - AChR vs Placebo - AChR; A Wilcoxon-Mann-Whitney Rank Sum Test of equality of change from baseline distributions between subjects diagnosed with MuSK-MG treated with amifampridine and placebo was conducted; Test type: Other; p = 0.2196, Wilcoxon (Mann-Whitney) — P-value for Wilcoxon-Mann-Whitney Test of Equality of change from baseline distributions between the amifampridine phosphate and placebo treatment groups

2. Secondary Outcome: Quantitative Myasthenia Gravis (QMG) Total Score Summary Statistics by Time Point and MG Type: Wilcoxon-Mann-Whitney Rank Sum Test Results
Description: Quantitative Myasthenia Gravis (QMG) assesses the patient's general body strength and fatigability. Each test item is scored on a scale of 0-3 with 3 representing the most severe symptom results and 0 representing no symptom results. Each item was assessed by the patient at Screening, the first (Day 1) and last day (Day 0) of the Run-in period and at the post-treatment visit. The post-treatment result will be the result obtained on Day 10. If the patient discontinued treatment early, the post-treatment result may be obtained at an earlier time point. The total QMG score was calculated as the sum of each item score, with a maximum score of 39 (most severe symptoms) and minimum score of 0 (least severe symptoms). The change from baseline (CFB) at Day 10 was assessed. A Wilcoxon-Mann-Whitney Rank Sum Test of equality of change from baseline distributions between subjects diagnosed with MuSK-MG treated with amifampridine and placebo was conducted.
Time Frame: Last day (Day 0) of the Run-in period and at the post-treatment visit (i.e., day 10 or the time at which a patient discontinued treatment early).
Population: The analysis of secondary outcome data was based on the Full Analysis Set population, which included all randomized patients who received at least one dose of study medication (amifampridine or placebo post randomization) and had at least one post-treatment efficacy assessment. Patients who discontinued with no post-randomization data (no Day 0 and no Day 10 data) were excluded from all efficacy analyses but were included in the safety analyses.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Amifampridine Phosphate - MuSK | Placebo - MuSK | Amifampridine Phosphate - AChR | Placebo - AChR
Number analyzed (Participants) | 27 | 28 | 7 | 8
Score on a Scale
  Baseline (Day 0) QMG Total Raw Score | 10.00 (3.873) | 8.64 (3.744) | 10.57 (3.359) | 14.13 (4.155)
  Post-Baseline (day 10 or time at which a patient discontinued treatment early) QMG Total Raw Score | 11.19 (5.367) | 10.16 (3.648) | 10.86 (3.024) | 14.43 (3.952)
  CFB QMG Total Score | 1.19 (3.99) | 1.80 (3.948) | 0.29 (3.039) | 0.86 (2.673)
Statistical Analysis 1: Comparison: Amifampridine Phosphate - MuSK vs Placebo - MuSK vs Amifampridine Phosphate - AChR vs Placebo - AChR; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3736, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were recorded for each patient from the time informed consent was obtained at Screening and continues through four weeks after the last dose or at the early discontinuation visit, for a total of approximately 52 days. Non-serious AEs were recorded for each patient after the first administration of study drug through the last visit or at the early discontinuation visit, for a total of approximately 10 days.
Description: Serious classification based on the FDA regulatory definition of a serious AE.
Groups:
- Amifampridine Phosphate: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day.
  The AEs reported within this treatment arm are those experienced by all participants who received Amifampridine Phosphate at the time of onset of the AE. Because this study has a run-in period where all subjects received Amifampridine Phosphate, the number of at-risk subjects in this treatment arm is identical to the overall number of at-risk participants. That is, the at-risk count includes those randomized to the Amifampridine Phosphate-Placebo sequence, Placebo - Amifampridine Phosphate sequence and those that received Amifampridine Phosphate during the open-label Run-in period but were not randomized for the crossover portion of the study.
- Placebo: Placebo Oral Tablet: tablets matching amifampridine phosphate, 3 to 4 times a day
  The AEs reported within this treatment arm are those experienced by participants who received Placebo at the time of onset of the AE. This includes those randomized to the Placebo - Amifampridine Phosphate sequence.
- Overall: Includes all participants who received study drug, including Amifampridine Phosphate during the open-label Run-in period or double-blind treatment period or Placebo during the double-blind treatment period.
Arm/Group | Amifampridine Phosphate | Placebo | Overall
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/36 | 0/86
Serious Adverse Events (participants affected / at risk) | 2/86 | 0/36 | 2/86
Other Adverse Events (participants affected / at risk) | 80/86 | 7/36 | 80/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine Phosphate (N=86) | Placebo (N=36) | Overall (N=86)
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 1
Myasthenia gravis crisis (Nervous system disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine Phosphate (N=86) | Placebo (N=36) | Overall (N=86)
Abdominal discomfort (Gastrointestinal disorders) | 5 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 12 | 0 | 12
Dyspepsia (Gastrointestinal disorders) | 7 | 0 | 7
Hypoaesthesia oral (Gastrointestinal disorders) | 9 | 0 | 9
Nausea (Gastrointestinal disorders) | 14 | 0 | 14
Paraesthesia oral (Gastrointestinal disorders) | 37 | 0 | 37
Fatigue (General disorders) | 10 | 2 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
Dizziness (Nervous system disorders) | 8 | 0 | 8
Headache (Nervous system disorders) | 11 | 0 | 11
Paraesthesia (Nervous system disorders) | 34 | 0 | 34
Peripheral coldness (Vascular disorders) | 5 | 0 | 5
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 3
Diplopia (Eye disorders) | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Asthenia (General disorders) | 3 | 0 | 3
Feeling cold (General disorders) | 3 | 0 | 3
Feeling hot (General disorders) | 2 | 0 | 2
Ear infection (Infections and infestations) | 2 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3
Sinusitis (Infections and infestations) | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 4
Myasthenia gravis (Nervous system disorders) | 1 | 1 | 2
Sensory disturbance (Nervous system disorders) | 3 | 0 | 3
Speech disorder (Nervous system disorders) | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Palpitations (Cardiac disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03304054/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03304054/SAP_001.pdf